CLINICAL TRIAL: NCT07136532
Title: Prediction of Fluid Responsiveness in Paediatric Patients With Septic Shock Using Carotid Doppler Ultrasonography and Echocardiography
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MD07/2024/2025
Record Dates: First submitted 2025-06-29; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-05

CONDITIONS: Septic Shock; Echocardiography Guided Fluid Management
Keywords: pediatric septic shock; echocardiography; carotid doppler
MeSH Terms: conditions — Shock, Septic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric patients with septic shock: All patients admitted at Paediatric Intensive care unit (PICU) during the period of the study and met the inclusion criteria.
  * Sex: Both males and females.
  * Age: 1 month to 16 years.
  * Sample size: 50 patients with septic shock admitted at PICU. All patients included in the study will be evaluated clinically and radiologically at fluid resuscitative phase of septic shock after fluid resuscitation.
  This evaluation will include:
  • Clinical examination:
  Clinical evaluation will be done initially and after fluid resuscitation:
  * Vital data (systolic, diastolic, and mean blood pressure, heart rate, Temperature).
  * Urine output, capillary perfusion time, Central venous pressure (CVP).
  * Detailed physical examination • Investigations:
  A) Laboratory:
  * Complete blood count.
  * Venous blood gases.
  * C-reactive protein.
  * Kidney function tests.
  * Albumin.
  * Serum lactate. -Echocardiography (measurement of stroke volume, stroke volume index,cardiac index) _carotid doppler ultrasonography
  Interventions: Diagnostic Test: echocardiography

INTERVENTIONS:
Diagnostic Test: echocardiography — Echocardiography will be performed using the ultrasound system echocardiographic equipment (Siemens Advanced Clinical Ultrasound Systems Optimized Navigation (ACUSON) P500), carotid doppler ultrasonography (Carotid blood flow and Corrected flow time) by using the ultrasound system echocardiographic equipment (Siemens ACUSON P500) .
  Those measurements will be done at time zero and upon completion of fluid resuscitation .
  • Statistical Analysis: All data will be collected, tabulated, and statistically analysed using International Business Machines_Statistical Package for the Social Sciences (IBM SPSS) version 27.

SUMMARY:
The goal of this study is to evaluate the role of carotid Doppler and Echocardiography as a predictor of fluid responsiveness in paediatric patients with septic shock.

and To evaluate the diagnostic accuracy of Aortic peak velocity and velocity time integral (VTI)variation in patients with septic shock during their fluid resuscitation phase as a reliable predictor of fluid responsiveness.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the role of carotid Doppler and Echocardiography as a predictor of fluid responsiveness in paediatric patients with septic shock.

and To evaluate the diagnostic accuracy of Aortic peak velocity and VTI variation in patients with septic shock during their fluid resuscitation phase as a reliable predictor of fluid responsiveness.All patients included in the study will be evaluated clinically and radiologically at fluid resuscitative phase of septic shock after fluid resuscitation.

This evaluation will include:

• Clinical examination:

Clinical evaluation will be done initially and after fluid resuscitation:

* Vital data (systolic, diastolic, and mean blood pressure, heart rate, Temperature).
* Urine output, capillary perfusion time, Central venous pressure (CVP).
* Detailed physical examination (chest, heart, and abdomen). • Investigations:

A) Laboratory:

* Complete blood count.
* Venous blood gases.
* C-reactive protein.
* Kidney function tests.
* Albumin.
* Serum lactate.
* Fibrinogen
* Serum electrolytes.
* Fibrinogen to albumin ratio

B) Imaging:

Echocardiography (measurement of stroke volume, stroke volume index, cardiac index, systemic vascular resistance index, Aortic peak velocity and VTI variation,, inferior vena cava (IVC)collapsibility index and IVC distensibility index)

ELIGIBILITY:
Inclusion criteria :

* Children aged 1 month to 16 years.
* Patients with septic shock admitted at the PICU during their fluid resuscitative phase were included.Septic shock was diagnosed according to phoenix sepsis score 2024

  • Exclusion criteria:
* Acquired and congenital heart disease.
* Acquired and congenital renal disease.
* Vascular anomalies (e.g. arteriovenous malformation, aneurysm).
* Suspected intracranial hypertension.
* Skin lesions or bandages at the sites of ultrasound or echo-cardiography examinations.
* Anatomical anomalies of the neck.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: o All Patients with septic shock admitted at the PICU during their fluid resuscitative phase during study time will be included.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the role of carotid Doppler and Echocardiography as a predictor of fluid responsiveness in paediatric patients with septic shock. | one year
  we use carotid Doppler and Echocardiography to predict the fluid responsiveness in paediatric patients with septic shock.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university _faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liteplo AS, Schleifer J, Marill KA, Huang CK, Gouker SK, Ratanski D, Diamond E, Filbin MR, Shokoohi H. Carotid Ultrasound in Assessing Fluid Responsiveness in Patients with Hypotension and Suspected Sepsis. Shock. 2021 Sep 1;56(3):419-424. doi: 10.1097/SHK.0000000000001755. PMID 33577247